## Informed Consent for Participation in Research 03/21/19

**Project Title:** Recovery Initiation and Management after Overdose (RIMO) **Principal Investigator:** Christy K. Scott, Ph.D., Chestnut Health Systems, 221 W. Walton,

Chicago, IL, 60610, Phone: (312) 664-4321, Fax: 312-664-4324,

Email: cscott@chestnut.org

Why is Lighthouse Institute doing this study? To see if we can help get people with a heroin or opioid problem who have overdosed into treatment. We also want to see if that helps make their lives better.

What will happen? You will be interviewed at our research office for about 30 minutes today, 3, 6 and 9 months from today. You can say no if you do not want to answer any question. You will also be asked to give a urine sample for testing at each interview. You will be asked to give us phone numbers and addresses so we can stay in touch with you. You will be photographed once by project staff, and the photograph will be attached to your Locator Form. The photograph will help project staff verify that the person they are interviewing each time is in fact you and not someone else. This photograph is also used to identify and locate you for follow-up interview purposes, and it may be shown to individuals to help locate you. These individuals will only be told that the researchers are trying to locate you for a health study in which you have agreed to participate. At the end of the project and after all follow-up interviews have been completed, a member of the project team will destroy the photograph. Everyone will receive a brochure on how to get into medication-assisted treatment. Half will be randomly selected to get linkage assistance with getting into treatment. Both the interviews and linkage sessions are audio recorded for quality assurance. You can ask these to be turned off at any time.

**How is the study organized?** You will be placed into 1 of 2 groups. One group will only do interviews. The other group will do interviews and receive help getting into and staying in treatment during the 9 month study. You will receive \$25 in gift cards for completing each interview and providing a urine sample, . No matter if you are in group 1 or group 2, you can always go to treatment and community-based recovery support services as usual.

How will information about me be shared with others? Your name and other information about you like your date of birth will be taken out of your file before it is given to anyone else. Your information will not be made public in any way. We have a **Certificate of Confidentiality** from the National Institutes of Health. It means we cannot be "forced" to give out any information to anyone that tells them you are in this study. We would only share information about you if you tell us you are going to hurt yourself or others. We also would share with the appropriate authorities your information if you tell us about a time when you hurt an older person or if you hurt or left a child uncared for.

What risks am I taking? There is a chance that some information about you could be found out. This is not usually a problem. Staff people who work on these studies need to follow federal laws. The federal laws protect your information. The people who interview you know how to protect your information. They must follow the rules in the **Certificate of Confidentiality.** 

What if I want to quit the study? You may take yourself out of the study at any time. You must give a written note to the person who is in charge of the study. You will still be able to go to your usual treatment or recovery services. When you stay in this study and take part in the interview,

you are helping us better understand people with drug problems and obstacles they face. Your answers to questions are important and give us helpful ideas.

| I agree to take part in the study: The study questions. I understand that I can choose out of this study at any time. I can continue study. No one has made any promises about information related to the study will be prowhen my information is looked at for a recombe protected by federal laws. | not to answer any question and<br>e with my usual treatment even<br>out how the study will turn out. I<br>tected and kept private accordi | I that I can take myseli<br>if I am not in the<br>My personal<br>ng to federal law. |
|---|---|---|
| I hereby agree / do not agree (countries consent form. I have been given a conquestions or concerns, I can contact the macharge is Dr. Christy Scott (Phone: 312-66 cscott@chestnut.org). If I have questions a can contact the person in charge of protections. | by of the consent form. I unders<br>nain person in charge of the stu<br>64-4321, Fax: 312-274-5335, e-<br>about my rights as a person in t | tand that if I have<br>dy. The person in<br>mail:<br>this research study, I |
| Participant (please print) | Participant (signature) | Date |
| Witness (signature) | Date | |
| IneligibleRefused (Reason | : <u> </u> | ) |

This consent automatically expires 5 years from the date it is signed.